CLINICAL TRIAL: NCT00020943
Title: A Phase II Study Of Intensive Induction Chemotherapy Followed By Autologous Stem Cell Transplantation Plus Immunotherapy For Mantle Cell Lymphoma
Brief Title: Chemotherapy and Rituximab With Peripheral Stem Cell Transplantation in Treating Patients With Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-59909; U10CA031946 (NIH); CALGB-59909; CDR0000068732 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: stage I mantle cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Rituximab; Carmustine; Cyclophosphamide; Cytarabine; Doxorubicin; Etoposide; Leucovorin; Methotrexate; Prednisone; Vincristine; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemo/immuno/autolog transplant (Experimental): Intensive chemotherapy followed by autologous stem cell transplant and immunotherapy for mantle cell lymphoma
  Interventions: Biological: filgrastim; Biological: rituximab; Drug: carmustine; Drug: cyclophosphamide; Drug: cytarabine; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: leucovorin calcium; Drug: methotrexate; Drug: prednisone; Drug: vincristine sulfate; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim — 5 ug/kg subQ daily day 4 until ANC >10,000 (or ANC> 5000 2X)Tx 1, 2, 4 10 ug/kg subQ daily day 14 until completion of PBSC collection Tx 3
  Other Names: G-CSF
Biological: rituximab — 375 mg/sq m IV infusion at , or = 400 mg/hr day 1 Tx 1, 2, days 5 & 12 Tx 3, and weekly for 2 doses Tx 5
Drug: carmustine — 15 mg/kg IV infusion over 2 hours Day 6, Tx 4
Drug: cyclophosphamide — 2000 mg/sq m IV infusion over 2 hours Day 3, Tx 1 & 2 100 mg/kg IV infusion over 2 hours Day 2, Tx 4
Drug: cytarabine — 2000 mg/sq m IV infusion BID over 2 hours x 8 doses Days 1-4, Tx 3
  Other Names: ara-C
Drug: doxorubicin hydrochloride — 50 mg/sq m IVP Day 3, Tx 1& 2
Drug: etoposide — 40 mg/kg total dose continuous IV infusion over 96 hours Days 1-4, Tx 3
Drug: leucovorin calcium — 50 mg/sq m IV infusion q 6 hours x 3 doses after MTX, then 10 mg/sq m IV/PO q 6 hrs until MTX levels <0.05 uM, Tx 1 & 2
Drug: methotrexate — 300 mg/sq m IV infusion over 4 hrs Day 2 Tx 1 & 2
Drug: prednisone — 100 mg/sq m PO Days 3-7, Tx 1 & 2
Drug: vincristine sulfate — 1.4 mg/sq m IVP Day 3, Tx 1 & 2
Procedure: peripheral blood stem cell transplantation — Stem cells collected during Tx 3 will be transfused follwing chemotx in Tx 4

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining chemotherapy and rituximab with peripheral stem cell transplantation in treating patients who have mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the two-year progression-free survival of patients with mantle cell lymphoma treated with intensive chemotherapy and rituximab with autologous peripheral blood stem cell (PBSC) transplantation.
* Determine the complete and partial response rates of patients treated with this regimen.
* Determine the disease-free and overall survival of patients treated with this regimen.
* Determine the autologous immune reconstitution in patients treated with this regimen.
* Determine the feasibility of this regimen in this patient population.
* Determine whether treatment with rituximab during autologous PBSC transplantation reduces the amount of contaminating lymphoma in the autologous PBSC product.

OUTLINE: This is a multicenter study.

Patients receive induction therapy comprising rituximab IV over 4-6 hours on day 1; methotrexate IV over 4 hours on day 2; cyclophosphamide IV over 2 hours, doxorubicin IV, and vincristine IV on day 3; and oral prednisone on days 3-7. Patients also receive leucovorin calcium IV every 6 hours beginning on day 3 and continuing until blood levels of methotrexate are safe. Filgrastim (G-CSF) is administered subcutaneously (SC) beginning on day 4 and continuing until blood counts recover.

Induction therapy repeats every 21-28 days for 2 courses in the absence of disease progression or unacceptable toxicity. Rituximab may be omitted during course 1 if circulating mantle cells are excessive. Patients may receive a third course if more than 15% persistent bone marrow involvement is documented.

Patients with stable or responding disease begin consolidation therapy 29 days after the start of the final course of induction therapy. Patients receive cytarabine IV over 2 hours twice daily and etoposide IV over 96 hours on days 1-4. Patients also receive rituximab IV over 4-6 hours on days 5 or 6 and 12 or 13 and G-CSF SC beginning on day 14 and continuing until leukapheresis is complete. Patients undergo leukapheresis beginning between days 22-25 and continuing until adequate CD34 cells are collected.

Beginning 4 weeks after recovery from consolidation therapy, patients receive high-dose therapy comprising carmustine IV over 2 hours on day -6, etoposide IV over 4 hours on day -4, and cyclophosphamide IV over 2 hours on day -2. Patients undergo autologous peripheral blood stem cell (PBSC) transplantation on day 0. Patients receive G-CSF SC beginning on day 6 and continuing until blood counts recover.

After blood counts recover and more than 35 days after autologous PBSC transplantation, patients receive rituximab IV over 4-6 hours weekly for 2 weeks.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually for up to 10 years.

PROJECTED ACCRUAL: At least 45 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed mantle cell lymphoma
* Presenting with at least one of the following:

  * Coexpression of CD20 (or CD19) and CD5 and a lack of CD23 expression by immunophenotyping
  * Positive for cyclin D1 by immunostaining
  * Presence of t(11,14) by cytogenetic analysis
  * Molecular evidence of bcl-1/IgH rearrangement
* Stage I-IV disease

  * Stage III or IV if nodular histology mantle cell lymphoma present
  * Any stage for other mantle cell histologies
  * No mantle zone histology
* No active CNS disease

  * No symptomatic meningeal lymphoma
  * No known CNS parenchymal lymphoma
  * Lumbar puncture showing mantle cell lymphoma allowed
* Bidimensionally measurable disease greater than 1 cm

  * Nonmeasurable disease includes the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
    * Lesions in a previously irradiated area

PATIENT CHARACTERISTICS:

Age:

* 18 to 69

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Hepatitis B surface antigen and hepatitis C antibody positive patients must meet all of the following criteria:

  * Bilirubin no greater than 2 times upper limit of normal (ULN)
  * AST no greater than 3 times ULN
  * Liver biopsy shows no greater than grade 2 fibrosis and no cirrhosis

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* LVEF at least 45% by MUGA or echocardiogram

Other:

* No known hypersensitivity to murine products
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No more than 1 prior dose of rituximab

Chemotherapy:

* No more than 1 prior cycle of chemotherapy
* At least 3 weeks since prior chemotherapy
* No other concurrent chemotherapeutic agents

Endocrine therapy:

* No chronic use of oral corticosteroids for ongoing medical condition
* No concurrent hormonal therapy except for non-lymphoma-related conditions (e.g., insulin for diabetes)
* Other concurrent corticosteroids for adrenal failure, diffuse alveolar hemorrhage, carmustine pneumonitis, or as an anti-emetic allowed

Radiotherapy:

* No prior radiotherapy for mantle cell lymphoma
* Concurrent palliative radiotherapy allowed
* Concurrent cranial radiotherapy for asymptomatic meningeal lymphoma allowed

Surgery:

* At least 2 weeks since prior major surgery

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2001-06; Primary Completion 2006-12 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years

SECONDARY OUTCOMES:
Response | 2 years
Survival | 5 years
  Disease free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Lloyd Damon, MD, Study Chair — University of California, San Francisco
Locations (81):
- United States (80):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Cedars-Sinai Comprehensive Cancer Center at Cedars-Sinai Medical Center, Los Angeles, California
  - Naval Medical Center - San Diego, San Diego, California
  - Veterans Affairs Medical Center - San Diego, San Diego, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Hematology/Oncology Faculty Practice, San Francisco, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Memorial Regional Cancer Center at Memorial Regional Hospital, Hollywood, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Fort Wayne Medical Oncology and Hematology, Incorporated, Fort Wayne, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - Las Vegas, Las Vegas, Nevada
  - New Hampshire Oncology-Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - University Hospital at State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Veterans Affairs Medical Center - Asheville, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - NorthEast Oncology Associates - Concord, Concord, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cape Fear Valley Health System, Fayetteville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Lenoir Memorial Hospital Cancer Center, Kinston, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital at Ohio State University, Columbus, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Veterans Affairs Medical Center - Dallas, Dallas, Texas
  - Green Mountain Oncology Group, Bennington, Vermont
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Incorporated - Roanoke, Roanoke, Virginia
  - St. Mary's Medical Center, Huntington, West Virginia
- Puerto Rico Cancer Center at University of Puerto Rico - Medical Sciences Campus, San Juan, Puerto Rico

REFERENCES:
- [Result] Damon LE, Johnson JL, Niedzwiecki D, Cheson BD, Hurd DD, Bartlett NL, Lacasce AS, Blum KA, Byrd JC, Kelly M, Stock W, Linker CA, Canellos GP. Immunochemotherapy and autologous stem-cell transplantation for untreated patients with mantle-cell lymphoma: CALGB 59909. J Clin Oncol. 2009 Dec 20;27(36):6101-8. doi: 10.1200/JCO.2009.22.2554. Epub 2009 Nov 16. PMID 19917845
- [Result] Hsi ED, Jung SH, Lai R, Johnson JL, Cook JR, Jones D, Devos S, Cheson BD, Damon LE, Said J. Ki67 and PIM1 expression predict outcome in mantle cell lymphoma treated with high dose therapy, stem cell transplantation and rituximab: a Cancer and Leukemia Group B 59909 correlative science study. Leuk Lymphoma. 2008 Nov;49(11):2081-90. doi: 10.1080/10428190802419640. PMID 19021050
- [Result] Damon LE, Johnson J, Niedzwiecki D, et al.: Immuno-chemotherapy (IC) and autologous stem cell transplant (ASCT) for untreated patients (pts) with mantle cell lymphoma (MCL): CALGB 59909. [Abstract] Blood 108 (11): A-2737, 2006.
- [Derived] Liu H, Johnson JL, Koval G, Malnassy G, Sher D, Damon LE, Hsi ED, Bucci DM, Linker CA, Cheson BD, Stock W. Detection of minimal residual disease following induction immunochemotherapy predicts progression free survival in mantle cell lymphoma: final results of CALGB 59909. Haematologica. 2012 Apr;97(4):579-85. doi: 10.3324/haematol.2011.050203. Epub 2011 Nov 18. PMID 22102709